CLINICAL TRIAL: NCT01326065
Title: Implementation of Laparoscopy-assisted Surgery for Colon Cancer. A Prospective Population-based Study
Brief Title: Implementation of Laparoscopy-assisted Surgery for Colon Cancer
Status: Terminated | Type: Observational
Why Stopped: Study had to be terminated due to lack of funding
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: SUH424503
Record Dates: First submitted 2011-02-27; First posted 2011-03-30 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to study the implementation of laparoscopy-assisted surgery for cure of colon cancer in daily surgical practice.

DETAILED DESCRIPTION:
Prospective observational study of laparoscopy-assisted surgery for resectable colon cancer with regard to short term and long term outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years
* diagnosis of colon cancer either endoscopically, radiologically or histologically proven
* No evidence of disseminated disease on CT scan
* T1-3 according to preoperative CT scan
* written informed consent to participate

Exclusion Criteria:

* preoperative diagnosis of locally advanced tumor (T4)
* suspicion of pathological lymph nodes outside anticipated resection area
* contraindications against laparoscopic surgery, e.g. known bowel adhesions, anesthesiological concerns
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients submitted for curative resection of colon cancer to the Dept. of Surgery, Stavanger University Hospital. Catchment area of the hospital consists of a population of 300.000 inhabitants, with Stavanger UH as the only institution with surgical service
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Long term outcome | 5 years
  overall survival and cancer specific survival, time to relapse

SECONDARY OUTCOMES:
Complications related to the surgical procedure | 30 days
  Anastomotic leaks; intra-abdominal infections; extra-abdominal complications, i.e. non-surgical site infections, cardiovascular events, death within 30 days after surgery
Quality of life | 1 year
  Quality of life as assessed by SF-36 questionary
Quality of the surgical specimen | 14 days
  R0 resection or not; number of lymph nodes harvested

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig Kørner, MD PhD, Principal Investigator — Helse Stavanger HF; Jens Christian Knapp, MD, Study Chair — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No